CLINICAL TRIAL: NCT01630239
Title: Technical Success, Safety, and Short-term Efficacy for MR-Guided Laser Ablation of Hepatic Tumors
Brief Title: MR-Guided Laser Ablation of Hepatic Tumors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Woodrum, Assistant Professor of Radiology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-000864
Record Dates: First submitted 2012-06-22; First posted 2012-06-28 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Soft Tissue Tumors
MeSH Terms: conditions — Soft Tissue Neoplasms | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Visualise Thermal Therapy System (Experimental)
  Interventions: Procedure: Laser ablation

INTERVENTIONS:
Procedure: Laser ablation — Laser ablation of hepatic tumors

SUMMARY:
This is a pilot study to investigate the performance of MR-guided Laser Induced Thermal Therapy (LITT) in the treatment of liver tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with soft tissue tumor metastases to the liver who are referred to Interventional Radiology for treatment.
* Surgery is not a viable or desirable alternative therapy at the time of enrollment
* Radiation therapy has failed or not indicated or can be safely postponed
* Tumor size ≤ 5 cm at its largest diameter
* Tumor position is not in the central liver hilum
* Performance status is ECOG 2 or better in adults
* Patient is able to undergo MRI

Exclusion Criteria:

* Patients with pacemaker or defibrillator
* Patients with metallic surgical clips close to the site of the intended ablation
* Pregnant women
* Patients with hilar liver lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
MR Images | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Woodrum, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States